CLINICAL TRIAL: NCT06162520
Title: Congenital Biliary Dilatation Diagnosis Based on 3D Morphological Characteristics
Status: Completed | Type: Observational
Sponsor: Tsinghua University (Other)
Collaborators: Beijing Tsinghua Chang Gung Hospital (Other)
Responsible Party: Principal Investigator, Jiaqi Dou, Principal Investigator, Tsinghua University
Other Study IDs: 21445-4-01
Record Dates: First submitted 2023-11-29; First posted 2023-12-08 (Actual); Last update posted 2023-12-08 (Actual); Status verified 2023-12

CONDITIONS: Congenital Biliary Dilatation
MeSH Terms: conditions — Choledochal Cyst

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Congenital biliary dilatation: Patients with congenital biliary dilatation diagnosed according to the Japanese Study Group on Congenital Biliary Dilatation (JSCBD) guideline.
  Interventions: Other: Contrast-enhanced computed tomography (CECT) and 3D morphological analysis
- Secondary biliary dilatation: Patients with secondary biliary dilatation attributed to choledocholithiasis or malignancies (hilar cholangiocarcinoma, pancreatic carcinoma, and distal cholangiocarcinoma).
  Interventions: Other: Contrast-enhanced computed tomography (CECT) and 3D morphological analysis

INTERVENTIONS:
Other: Contrast-enhanced computed tomography (CECT) and 3D morphological analysis — Diagnosis models are established using quantitative morphological characteristics extracted from the 3D reconstructed bile duct from contrast-enhanced computed tomography (CECT) images.

SUMMARY:
Congenital biliary dilatation necessitates timely intervention owing to potential complications. This study endeavors to enhance diagnostic precision using quantitative three-dimensional morphological characteristics. Objectives involve developing models to differentiate congenital from secondary biliary dilatation and identify intrahepatic involvement. Employing machine learning, robust diagnostic models aim to elevate clinical detection rates and improve accuracy.

DETAILED DESCRIPTION:
Congenital biliary dilatation is a primary anomaly affecting the biliary tract. It can involve the extrahepatic bile ducts, intrahepatic bile ducts, or the entire biliary system, including the common bile duct. Patients with congenital biliary dilatation exhibit abnormal expansion of the bile duct system, which can lead to complications such as bile duct stones, pancreatic inflammation, and even bile duct cancer. Timely and accurate diagnosis, followed by surgical intervention to remove the dilated bile duct lesion, is crucial for the treatment of choledochal dilation. However, the differentiation of congenital biliary dilatation in clinical practice poses challenges, primarily due to the limitations of subjective physician experience and macroscopic imaging features, making it difficult to achieve high sensitivity in discerning congenital biliary dilatation. Particularly, in distinguishing between congenital biliary dilatation and secondary biliary dilatation, the similarities of the bile ducts limit the precision of clinical decisions. Therefore, this study aims to address the current challenges in the differential diagnosis of congenital biliary dilatation and secondary biliary dilatation by quantitatively describing the morphology of dilated bile ducts. Moreover, this study plans to build a predictive model of intrahepatic bile duct dilatation to provide more comprehensive clinical support. Specifically, the research objectives are outlined as follows:

1. Establish a diagnostic model for congenital biliary dilatation utilizing three-dimensional morphological characteristics, especially quantitative shape- and diameter-based characteristics, to enhance the accurate discrimination between congenital biliary dilatation and secondary biliary dilatation.
2. Develop a model for identifying intrahepatic involvement of congenital biliary dilatation, aiming to provide more precise information for surgical planning and supportive treatment.
3. Construct robust diagnostic models using machine learning with quantitative three-dimensional morphological characteristics, aiming to increase clinical detection rates and accuracy, thereby achieving risk stratification for patients with biliary dilatation.

ELIGIBILITY:
Inclusion Criteria:

* The patients with biliary dilation who underwent contrast-enhanced computed tomography (CECT) at Beijing Tsinghua Chang Gung Hospital from 2014 to 2022.

Exclusion Criteria:

* Patients without pre-operative CECT scans or developing cholangiocarcinoma due to congenital biliary dilatation.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with congenital biliary dilatation diagnosed according to the Japanese Study Group on Congenital Biliary Dilatation (JSCBD) guideline or secondary bile duct dilatation due to choledocholithiasis or malignancies such as hilar cholangiocarcinoma, pancreatic carcinoma, and distal cholangiocarcinoma who underwent contrast-enhanced computed tomography (CECT) at Beijing Tsinghua Chang Gung Hospital from 2014 to 2022.
Sampling Method: Non-Probability Sample
Enrollment: 550 (Actual)
Dates: Start 2021-12-17 (Actual); Primary Completion 2022-12-16 (Actual); Study Completion 2022-12-16 (Actual)

PRIMARY OUTCOMES:
Area under the Receiver Operating Characteristic curve (AUROC) of the diagnostic models for the differential diagnosis of congenital and secondary biliary dilatation and the identification of intrahepatic involvement | Pre-operation
  The area under the ROC curve is calculated by integrating the ROC curve, which plots Sensitivity against 1 - Specificity.

SECONDARY OUTCOMES:
Area under the Precision-Recall curve (AUPRC) of the diagnostic models for the differential diagnosis of congenital and secondary biliary dilatation and the identification of intrahepatic involvement | Pre-operation
  The area under the precision-recall curve is determined by integrating the Precision-Recall curve, which plots Precision against Recall.
Sensitivity of the diagnostic models for the differential diagnosis of congenital and secondary biliary dilatation and the identification of intrahepatic involvement | Pre-operation
  Sensitivity is calculated as the ratio of true positives to the sum of true positives and false negatives.
Specificity of the diagnostic models for the differential diagnosis of congenital and secondary biliary dilatation and the identification of intrahepatic involvement | Pre-operation
  Specificity is calculated as the ratio of true negatives to the sum of true negatives and false positives.
Accuracy of the diagnostic models for the differential diagnosis of congenital and secondary biliary dilatation and the identification of intrahepatic involvement | Pre-operation
  Accuracy is calculated as the ratio of the sum of true positives and true negatives to the total number of cases.

CONTACTS AND LOCATIONS:
Overall Officials: Huijun Chen, Ph.D., Study Director — Tsinghua University; Jiahong Dong, M.D., Study Chair — Beijing Tsinghua Chang Gung Hospital
Locations (1):
- Beijing Tsinghua Chang Gung Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ishibashi H, Shimada M, Kamisawa T, Fujii H, Hamada Y, Kubota M, Urushihara N, Endo I, Nio M, Taguchi T, Ando H; Japanese Study Group on Congenital Biliary Dilatation (JSCBD). Japanese clinical practice guidelines for congenital biliary dilatation. J Hepatobiliary Pancreat Sci. 2017 Jan;24(1):1-16. doi: 10.1002/jhbp.415. Epub 2017 Jan 22. PMID 28111910
- [Derived] Dou J, Jiang N, Zeng J, Wang S, Tian S, Shan S, Li Y, Xu Z, Lin X, Jin S, Dong J, Chen H. Novel 3D morphological characteristics for congenital biliary dilatation diagnosis: a case-control study. Int J Surg. 2024 May 1;110(5):2614-2624. doi: 10.1097/JS9.0000000000001204. PMID 38376858